CLINICAL TRIAL: NCT00347841
Title: Efficacy of Bimatoprost 0.03% in Patients Who Are Low-Responders to Latanoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 5178
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost; Latanoprost

INTERVENTIONS:
Drug: Bimatoprost 0.03%, Latanoprost

SUMMARY:
To evaluate the IOP-lowering efficacy of bimatoprost 0.03% in patients found to be low-responders to latanoprost therapy.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age

  * Documented low-responder to latanoprost therapy as delineated in the outline above.
  * Diagnosis of open-angle glaucoma or ocular hypertension
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication to bimatoprost or any component of any study medication

  * Uncontrolled systemic disease
  * Active ocular disease other than glaucoma or ocular hypertension
  * Required use of ocular medications other than the study medications during the study (intermittent use of artificial tear solutions will be permitted)
  * History of intraocular surgery within the last 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noecker, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- Dr. Noecker, Pittsburgh, Pennsylvania, United States